CLINICAL TRIAL: NCT01833468
Title: FUNCTIONAL LIMITATIONS DUE TO the FOOT INVOLVEMENT IN SPONDYLOARTHRITIS
Status: Completed | Type: Observational
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Foot-SpA
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: ankylosing spondylitis; Psoriatic arthritis; Foot; FAOS; SpA-TRI
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Seronegative spondyloarthritis (SpA) is a group of rheumatic diseases Foot involvement of the SpA is common and enthesitis, erosive changes or ankylosis are the frequent lesions. The functional status of the SpA patients are usually evaluated globally.The aim of this study is to assess specifically the foot -related functional limitations of the SpA patients.

DETAILED DESCRIPTION:
SpA patients who had foot pain at least for 4 weeks and those having bilateral anteroposterior and lateral feet x-rays will be included into the study. Foot x-rays will be evaluated by a radiologist by using the spondyloarthropathy tarsal radiographic index (SpA-TRI). The foot related functional status of the patients will be determined by the Turkish version of the Foot and Ankle Outcome Score (FAOS).

ELIGIBILITY:
Inclusion Criteria:

* SpA patients who had foot pain at least for 4 weeks
* Those having bilateral anteroposterior and lateral feet x-rays will be included into the study

Exclusion Criteria:

* Patients who had flatfoot
* Previous foot surgery
* Any other disorder unrelated to the SpA will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with SpA and foot pain
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The foot-related functional status of SpA patients | 1 month
  The foot related functional status of the subjects will be measured with Foot Ankle Outcome Score (FAOS)

CONTACTS AND LOCATIONS:
Overall Officials: nihal ozaras, ass.prof, Principal Investigator — Bezmialem Vakif University